CLINICAL TRIAL: NCT02601989
Title: Effects on Insulin Resistance With the Phosphodiesterase-5 Inhibitor Tadalafil in Type 2 Diabetes - a Double-blind, Placebo-controlled Crossover Study
Brief Title: Effects on Insulin Resistance With Tadalafil in Type 2 Diabetes - a Double-blind, Placebo-controlled Crossover Study
Acronym: MAKROTAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2015-09-14; 2015-000573-12 (EudraCT Number)
Record Dates: First submitted 2015-10-26; First posted 2015-11-11 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tadalafil (Experimental): Per oral intake of tadalafil 20 mg o.d. for six weeks
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator): Per oral intake of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil
  Arms: Tadalafil
Drug: Placebo — Per oral intake of placebo for six weeks
  Arms: Placebo

SUMMARY:
The aim is to continue our program on PDE5 inhibition by evaluating effects on insulin resistance, including glucose metabolism and subclinical inflammation, after a 6-week administration of tadalafil in T2D patients. The primary objective is to study the effect of tadalafil compared with placebo on insulin sensitivity during a euglycemic hyperinsulinemic clamp.

This is a double-blind, placebo-controlled crossover study with one study site. Twenty-five T2D patients will be recruited and randomized to per oral intake of tadalafil 20 mg o.d. for six weeks and after a wash-out period of eight weeks intake of placebo for another six weeks, or vice versa. At the end of each 6 week treatment period a glucose clamp, subcutaneous needle biopsies as well as muscle and subcutaneous microdialysis will be performed. Endothelial function tests and arginin stimulation of insulin secretion tests will be performed after 3 weeks in each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. T2D patient, previously diagnosed by fasting or 2-hr OGTT plasma glucose levels
2. Age females: 55-70 yrs (post-menopausal state defined as natural amenorrhea for at least 12 months); Age males: 40-70 yrs
3. BMI: 27-40 kg/m2
4. HbA1c < 60 mmol/mol
5. Type 2 diabetes duration > 3 months and < 10 yrs
6. Understand and speak Swedish

Exclusion Criteria:

1. Diabetes treatment with glitazones, GLP-1 analogues or DPP-IV inhibitors
2. Anti-hypertensive therapy with beta-blockers, ACE-inhibitors and/or angiotensin-II receptor blockers
3. Significant microvascular complications e.g. nephropathy (GFR<60), proliferative retinopathy and symptomatic neuropathy e.g. postural hypotension
4. Previous significant vascular disease including angina pectoris and myocardial infarction, cerebral artery disease e.g. history of transient ischemic attacks and peripheral artery disease with no palpable pulses
5. Smoking > 10 cig/day and/or smokeless tobacco > one can per 2 days
6. Concurrent use of nitrates or NO donors, or an apparent risk that there may be a need of such medication
7. Cardiac failure (stages NYHA II-IV)
8. Uncontrolled hypertension > 170/105 mm Hg
9. Apparent ECG-pathology indicating current or previous myocardial ischemia;
10. Males with erectile dysfunction
11. Hemophilia or a history of bruises or hepatic failure (> 2-fold increase upper limit normal values of ASAT/ALAT)
12. Hypotension
13. Treatment with doxazosin
14. Anything in the contact with the patient that makes the doctor to believe that he/she will be uncompliant to the protocol.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity | 6 week treatment with drug or placebo
  To evaluate the effect (difference in glucose disposal rate (mg/kg/min)) of daily administration of 20 mg tadalafil for 6 weeks ("chronic" treatment) on insulin sensitivity in muscle by assessing glucose disposal rate during a 3-hour euglycemic hyperinsulinemic glucose clamp (120 mU/m2/min) in T2D patients

SECONDARY OUTCOMES:
Mean glucose (HbA1c, mmol/mol) in blood | Up to 6 weeks after start of treatment.
  Evaluation the effect of chronic tadalafil treatment on glucose metabolism and beta-cell function as measured by mean blood glucose (HbA1c)
Fasting plasma glucose levels (mmol/l) | Up to 6 weeks after start of treatment.
  Evaluation the effect of chronic tadalafil treatment on glucose metabolism and beta-cell function as measured by circulating glucose levels
Arginine-induced insulin secretion (area under curve, AUC, mU/l/min) in blood | 3 weeks after start of treatment.
  Glucose metabolism and beta-cell function as measured by arginine-induced insulin secretion (difference in AUC, mU/l/min).
Levels interstitial insulin | Up to 6 weeks after start of treatment.
  levels interstitial insulin (mU/l)
Lactate concentrations in insulin sensitive tissues | Up to 6 weeks after start of treatment.
  Lactate concentrations (micromoles/l) in insulin sensitive tissues
Levels of inflammatory markers in blood | Up to 6 weeks after start of treatment.
  Difference in endothelin-1 levels (pg/ml)
Endothelial function in peripheral arteries measured with EndoPAT, measured as difference in reactive hyperemia | 3 weeks after start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Per-Anders Jansson, MD, Principal Investigator — Göteborg University
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Fryk E, Rodrigues Silva VR, Bauza-Thorbrugge M, Schmelz M, Gan LM, Strindberg L, Jansson PA. Feasibility of high-dose tadalafil and effects on insulin resistance in well-controlled patients with type 2 diabetes (MAKROTAD): a single-centre, double-blind, randomised, placebo-controlled, cross-over phase 2 trial. EClinicalMedicine. 2023 May 4;59:101985. doi: 10.1016/j.eclinm.2023.101985. eCollection 2023 May. PMID 37256099